CLINICAL TRIAL: NCT06243445
Title: Transthoracic Echocardiography With Bubble Test for Tip Location of Central Venous Catheters: a "Push to Bubble" Time Analysis
Brief Title: Echocardiography With Bubble Test for Tip Location of Central Venous Catheters
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Dr.ssa Gabriella Arlotta, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5762
Record Dates: First submitted 2024-01-28; First posted 2024-02-06 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Surgery Patient
Keywords: central venous catheter tip location; transthoracic echocardiography; bubble test
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients underwent cardiac surgery with need for a central venous catheter: Patients underwent cardiac surgery with need for a central venous catheter and indication to intraoperative trans esophageal echocardiography
  Interventions: Diagnostic Test: Transthoracic echocardiography for central venous catheter tip location

INTERVENTIONS:
Diagnostic Test: Transthoracic echocardiography for central venous catheter tip location — Measure of time between injection of echographic contrast in the distal lumen of a central venous catheter, inserted via supra/infra clavicular right veins, and visualization, using transthoracic echocardiography, of micro bubbles in right atrium with the catheter tip positioned under transesophageal ultrasound control in four different positions: right atrium, cavo-atrial junction (CAJ), at 4 centimeters proximal to CAJ, in superior vena cava and at 8 centimeters proximal to CAJ

SUMMARY:
The goal of this prospective observational study is to test the accuracy of the transthoracic echocardiography with bubble test to verify the location of the tip of the central venous catheter in patients undergoing cardiac surgery procedures. The main questions it aims to answer are:

1. Is there a difference in time elapsed between the injection of a saline solution (echogenic contrast) through a central venous catheter and the visualization of micro bubbles in right atrium ("push to bubbles" time) with transthoracic echocardiography, when the catheter tip is placed in four different positions identified by transesophageal echocardiography?
2. Is there a difference in time for the right atrium to be completely filled by bubbles after saline injection in a central venous catheter with the tip placed in four different positions identified by transesophageal echocardiography?
3. In what percentage of patients the acoustic window is good enough to evaluate "push to bubbles" time?
4. Is there a difference in "push to bubbles" time between different echocardiographic projections?
5. Is the bubbles flow laminar or turbulent in the four different positions?
6. Is there a relation between "push to bubble" time and heart rate, blood pressure, pulmonary artery pressure, central venous pressure and cardiac output measured through a pulmonary artery catheter?

Participants will require simultaneously a central venous catheter and an intraoperative transesophageal echocardiography.

DETAILED DESCRIPTION:
The placement of central vascular access devices (VADs), with cervical-thoracic or femoral insertion (such as CICC, Central Inserted Central Catheter, and FICC, Femoral Inserted Central Catheter), as well as peripheral insertion (PICC, Peripherally Inserted Central Catheter), is a common procedure for patients admitted to the Intensive Care Unit and for patients undergoing major surgery or prolonged infusion therapy.

To reduce the incidence of complications related to improper positioning of the central venous catheter, the tip should be positioned in the lower part of the superior vena cava or in the upper part of the right atrium near the cavo-atrial junction, identified by the crista terminalis.

Among the methods used to verify the correct tip placement, the intracavitary ECG method is strongly recommended by various international guidelines, and its use has been widely validated in terms of safety, efficacy, and accuracy. However, the intracavitary ECG method, based on the principle that the appearance of a high P-wave indicates the proximity of the tip to the cavo-atrial junction, has limitations when it comes to patients with non-sinus rhythm. Recent studies are validating the use of modified intracavitary ECG in patients with atrial fibrillation, but in other cases where a P-wave is not visible, the method is not applicable.

Various methods for ultrasound-guided placement and confirmation of the final tip position have been developed, also because the chest X-ray performed at the patient's bedside has proven to be a less accurate method due to the lack of definite findings of the cavo-atrial junction.

Transesophageal echocardiography (TEE), while being the method of choice as it allows direct visualization of the cavo-atrial junction and, therefore, the real position of both the guidewire and the tip of the catheter at the end of placement, remains an invasive method that is difficult to perform outside of cardiac operating rooms.

Transthoracic echocardiography may allow for the direct visualization of the tip of the VAD inside the heart chambers or indirectly assessing the tip's position by injecting echogenic contrast. Echogenic contrast refers to a rapid bolus of 5-20 ml of 0.9% saline solution, with or without the addition of 1 ml of air, vigorously shaken to create micro bubbles that can be easily visualized during the echocardiographic exam. The bolus is injected into the VAD once it has been positioned, and the micro bubbles are visualized in the right atrium, using transthoracic echocardiography. In nearly all studies, the VAD is considered in the correct position if the micro bubbles appear in the atrium within 2 seconds of injection ("push to bubble" time); otherwise, it is not considered correctly positioned if the bubbles appear after 2 seconds, but in one study, the adequate time was considered to be less than 500 ms. In almost all echocardiography studies, however, the reference method used to evaluate and confirm the VAD tip position has been chest radiography, which has been proven to be a less accurate method; moreover, literature shows significant variations in the indicative times for the visualization of micro bubbles that suggest incorrect position (range 0.5-2 seconds).

In this context, it could be useful to determine accurately if different "push to bubble" times are indicative for different positions of the VAD tip. For this purpose, the echogenic contrast (10 ml of 0,9% saline solution with the addition of 1 ml of air vigorously shaken to create micro bubbles) will be injected in the distal lumen of a VAD, whose tip is positioned in four different points, identified with using transesophageal echocardiography and the time from the contrast injection to the visualization of the bubbles in right atrium will be recorded using transthoracic echocardiography.

The four positions in which the catheter tip will be placed are: right atrium, cavo-atrial junction (CAJ), at 4 centimeters proximal to the CAJ in superior vena cava and at 8 centimeters to the CAJ. The catheter tip positions in right atrium and at CAJ will be directly evaluated using 2D and 3D transesophageal echocardiography, the other positions will be obtained moving the catheter back 4 and 8 centimeters from the CAJ. The transthoracic echocardiography will be carried out always by the same cardiologist trained in echocardiography unaware of the purpose of the study. The time measurements will be carried out always by the same cardiac anaesthesiologist, trained in echocardiography, unaware of the different catheter tip positions.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* written informed consent from the patient
* intra-operative need for a central venous catheterization via the supra/infra clavicular right veins (centrally inserted central catheter, CICC)
* indication to intra-operative Trans Esophageal Ultrasound (TEE) based on American Society of Anesthesiologists (ASA)

Exclusion Criteria:

* contraindications to TEE based on American Society of Anesthesiologists (ASA) recommendations (esophageal or gastric diseases or previous surgery)
* emergency procedures
* central VAD already placed
* need for a CICC via supra/infra clavicular left veins
* need for a femorally inserted central catheter (FICC)
* need for a peripherally inserted central catheter (PICC)
* tricuspid valve regurgitation
* hemodynamic instability/ presence of an intra-aortic ballon pump (IABP)
* absence of septal atrial defect

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll patients of both sexes, aged> 18 years, with cardiovascular disease, who must undergo cardiac surgery
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2025-11-27 (Actual)

PRIMARY OUTCOMES:
Difference in "push to bubbles" time recorded with the catheter tip placed in four different positions by three different ultrasound views; measure in position 1: right atrium, using subcostal 4-chamber view | Immediately after the induction of anesthesia, placement of transesophageal probe and insertion of a central venous catheter. The video recorded will be analyzed immediately after the end of the procedure
  After the insertion of a central venous catheter in the supraclavicular right area by ultrasound guidance and direct Seldinger technique, under transesophageal ultrasound control, the catheter tip will be placed in right atrium, 2 cm below the CAJ; the echographic contrast will be injected through the proximal end of the catheter connected, via an Arrow-Johans adapter (Teleflex) and a dedicated ECG cable (Teleflex), to the transthoracic ultrasound machine. The video with the micro bubbles injected will be recorded by a cardiologist expert in echocardiography, unaware of the purpose of the study, using a subcostal 4-chamber view. Later a cardiac anesthesiologist, unaware of the purpose of the position of the catheter, will measure the time elapsed between the first positive wave created by the contrast injection on the intracavitary ECG recorded by the transthoracic ultrasound machine and the time in which the bubbles will appear in the right atrium.
Difference in "push to bubbles" time recorded with the catheter tip placed in four different positions by three different ultrasound views; measure in position 1: right atrium, using subcostal bicaval view | Immediately after the video recorded with the catheter tip placed in right atrium using subcostal 4-chamber view
  With the procedure described above, the "push to bubble" time will be measured with the catheter tip placed in right atrium using subcostal bicaval view
Difference in "push to bubbles" time recorded with the catheter tip placed in four different positions by three different ultrasound views; measure in position 1: right atrium, using apical 4-chamber view | Immediately after the video recorded with the catheter tip placed in right atrium using subcostal bicaval view
  With the procedure described above, the "push to bubble" time will be measured with the catheter tip placed in right atrium using apical 4-chamber view
Difference in "push to bubbles" time recorded with the catheter tip placed in four different positions by three different ultrasound views; measure in position 2: cavo-atrial junction (CAJ), using subcostal 4-chamber view | Immediately after the video recorded with the catheter tip placed in right atrium using apical 4-chamber view
  With the procedure described above, the "push to bubble" time will be measured with the catheter tip placed at the CAJ, using subcostal 4-chamber view
Difference in "push to bubbles" time recorded with the catheter tip placed in four different positions by three different ultrasound views; measure in position 2: cavo-atrial junction (CAJ), using subcostal bicaval view | Immediately after the video recorded with the catheter tip placed at the CAJ using subcostal 4-chamber view
  With the procedure described above, the "push to bubble" time will be measured with the catheter tip placed at the CAJ, using subcostal bicaval view
Difference in "push to bubbles" time recorded with the catheter tip placed in four different positions by three different ultrasound views; measure in position 2: cavo-atrial junction (CAJ), using apical 4-chamber view | Immediately after the video recorded with the catheter tip placed at the CAJ using subcostal bicaval view
  With the procedure described above, the "push to bubble" time will be measured with the catheter tip placed at the CAJ, using apical 4-chamber view
Difference in "push to bubbles" time recorded with the catheter tip placed in four different positions by three different ultrasound views; measure in position 3: at 4 centimeters proximal to CAJ in superior vena cava, using subcostal 4-chamber view | Immediately after the video recorded with the catheter tip placed at the CAJ using apical 4-chamber view
  With the procedure described above, the "push to bubble" time will be measured with the catheter tip placed at , 4 centimeters proximal to CAJ in superior vena cava, using subcostal 4-chamber view
Difference in "push to bubbles" time recorded with the catheter tip placed in four different positions by three different ultrasound views; measure in position 3: at 4 centimeters proximal to CAJ in superior vena cava, using subcostal bicaval view | Immediately after the video recorded with the catheter tip at 4 centimeters proximal to CAJ, in superior vena cava, using subcostal 4-chamber view
  With the procedure described above, the "push to bubble" time will be measured with the catheter tip placed at 4 centimeters proximal to CAJ in superior vena cava, using subcostal bicaval view
Difference in "push to bubbles" time recorded with the catheter tip placed in four different positions by three different ultrasound views; measure in position 3: at 4 centimeters proximal to CAJ in superior vena cava, using apical 4-chamber view | Immediately after the video recorded with the catheter tip at 4 centimeters proximal to CAJ, in superior vena cava, using subcostal bicaval view
  With the procedure described above, the "push to bubble" time will be measured with the catheter tip placed at 4 centimeters proximal to CAJ in superior vena cava, using apical 4-chamber view
Difference in "push to bubbles" time recorded with the catheter tip placed in four different positions by three different ultrasound views; measure in position 4: at 8 centimeters proximal to CAJ, using subcostal 4-chamber view | Immediately after the video recorded with the catheter tip at 4 centimeters proximal to the CAJ, in superior vena cava, using apical 4-chamber view
  With the procedure described above, the "push to bubble" time will be measured with the catheter tip placed at 8 centimeters proximal to the CAJ, using subcostal 4-chamber view
Difference in "push to bubbles" time recorded with the catheter tip placed in four different positions by three different ultrasound views; measure in position 4: at 8 centimeters proximal to CAJ, using subcostal bicaval view | Immediately after the video recorded with the catheter tip at 8 centimeters, using subcostal 4-chamber view
  With the procedure described above, the "push to bubble" time will be measured with the catheter tip placed at 8 centimeters proximal to the CAJ, using subcostal bicaval view
Difference in "push to bubbles" time recorded with the catheter tip placed in four different positions by three different ultrasound views; measure in position 4: at 8 centimeters proximal to CAJ, using apical 4-chamber view | Immediately after the video recorded with the catheter tip at 8 centimeters, using subcostal bicaval view
  With the procedure described above, the "push to bubble" time will be measured with the catheter tip placed at 8 centimeters proximal to the CAJ, using apical 4-chamber view

SECONDARY OUTCOMES:
Difference in time for the right atrium to be completely filled by micro bubbles; measure with the catheter tip placed in position 1: right atrium, using subcostal 4-chamber view | Immediately after measuring "push to time" in the video recorded with the catheter tip in right atrium, using subcostal 4-chamber view
  The time needed for the right atrium to be completely filled by micro bubbles will be measured analyzing the video recorded with the catheter tip in right atrium using subcostal bicaval view
Difference in time for the right atrium to be completely filled by micro bubbles; measure with the catheter tip placed in position 1: right atrium, using subcostal bicaval view | Immediately after measuring "push to time" in the video recorded with the catheter tip placed in right atrium using subcostal bicaval view
  The time needed for the right atrium to be completely filled by micro bubbles will be measured analyzing the video recorded with the catheter tip in right atrium using subcostal bicaval view
Difference in time for the right atrium to be completely filled by micro bubbles; measure with the catheter tip placed in position 1: right atrium, using apical 4-chamber view | Immediately after measuring "push to time" in the video recorded with the catheter tip placed in right atrium, using apical 4-chamber view
  The time needed for the right atrium to be completely filled by micro bubbles will be measured analyzing the video recorded with the catheter tip in right atrium using apical 4-chamber view
Difference in time for the right atrium to be completely filled by micro bubbles; measure with the catheter tip placed in position 2: cavo-atrial junction (CAJ), using subcostal 4-chamber view | Immediately after measuring "push to time" in the video recorded with the catheter tip placed at cavo-atrial junction (CAJ), using subcostal 4-chamber view
  The time needed for the right atrium to be completely filled by micro bubbles will be measured analyzing the video recorded with the catheter tip placed at the CAJ, using subcostal 4-chamber view
Difference in time for the right atrium to be completely filled by micro bubbles; measure with the catheter tip placed in position 2: cavo-atrial junction (CAJ), using subcostal bicaval view | Immediately after measuring "push to time" in the video recorded with the catheter tip placed at cavo-atrial junction (CAJ), using subcostal bicaval
  The time needed for the right atrium to be completely filled by micro bubbles will be measured analyzing the video recorded with the catheter tip placed at the CAJ, using subcostal bicaval view
Difference in time for the right atrium to be completely filled by micro bubbles; measure with the catheter tip placed in position 2: cavo-atrial junction (CAJ), using apical 4-chamber view | Immediately after measuring "push to time" in the video recorded with the catheter tip placed at cavo-atrial junction (CAJ), using apical 4-chamber view
  The time needed for the right atrium to be completely filled by micro bubbles will be measured analyzing the video recorded with the catheter tip placed at the CAJ, using apical 4-chamber view
Difference in time for the right atrium to be completely filled by micro bubbles; measure with the catheter tip placed in position 3: 4 centimeters proximal to CAJ in superior vena cava, using subcostal 4-chamber view | Immediately after measuring "push to time" in the video recorded with the catheter tip placed at 4 centimeters proximal to CAJ in superior vena cava, using subcostal 4-chamber view
  The time needed for the right atrium to be completely filled by micro bubbles will be measured analyzing the video recorded with the catheter tip placed at 4 centimeters proximal to CAJ in superior vena cava, using subcostal 4-chamber view
Difference in time for the right atrium to be completely filled by micro bubbles; measure with the catheter tip placed in position 3: 4 centimeters proximal to CAJ in superior vena cava, using subcostal bicaval view | Immediately after measuring "push to time" in the video recorded with the catheter tip placed at 4 centimeters proximal to CAJ in superior vena cava, using subcostal bicaval view
  The time needed for the right atrium to be completely filled by micro bubbles will be measured analyzing the video recorded with the catheter tip placed at 4 centimeters proximal to CAJ using subcostal bicaval view
Difference in time for the right atrium to be completely filled by micro bubbles; measure with the catheter tip placed in position 3: 4 centimeters proximal to CAJ in superior vena cava, using apical 4-chamber view | Immediately after measuring "push to time" in the video recorded with the catheter tip placed at 4 centimeters proximal to CAJ in superior vena cava, using apical 4-chamber view
  The time needed for the right atrium to be completely filled by micro bubbles will be measured analyzing the video recorded with the catheter tip placed at 4 centimeters proximal to CAJ in superior vena cava, using apical 4-chamber view
Difference in time for the right atrium to be completely filled by micro bubbles; measure with the catheter tip placed in position 4: 8 centimeters proximal to CAJ, using subcostal 4-chamber view | Immediately after measuring "push to time" in the video recorded with the catheter tip placed at 8 centimeters proximal to CAJ, using subcostal 4-chamber view
  The time needed for the right atrium to be completely filled by micro bubbles will be measured analyzing the video recorded with the catheter tip placed at 8 centimeters proximal to the CAJ, using subcostal 4-chamber view
Difference in time for the right atrium to be completely filled by micro bubbles; measure with the catheter tip placed in position 4: 8 centimeters proximal to CAJ, using subcostal bicaval view | Immediately after measuring "push to time" in the video recorded with the catheter tip placed at 8 centimeters proximal to CAJ, using subcostal bicaval view
  The time needed for the right atrium to be completely filled by micro bubbles will be measured analyzing the video recorded with the catheter tip placed at 8 centimeters proximal to the CAJ, using subcostal bicaval view
Difference in time for the right atrium to be completely filled by micro bubbles; measure with the catheter tip placed in position 4: 8 centimeters proximal to CAJ, using apical 4-chamber view | Immediately after measuring "push to time" in the video recorded with the catheter tip placed at 8 centimeters proximal to CAJ, using apical 4-chamber view
  The time needed for the right atrium to be completely filled by micro bubbles will be measured analyzing the video recorded with the catheter tip placed at 8 centimeters proximal to the CAJ, using apical 4-chamber view
Percentage in which "push to bubbles" time is evaluable using subcostal 4-chamber view | Immediately after every patient recruited will be evaluated with ultrasound in subcostal 4-chamber view
  To measure the percentage of the patients in which acoustic window is good enough to evaluate "push to bubbles" time using subcostal 4-chamber view.
Percentage in which "push to bubbles" time is evaluable using subcostal bicaval view | Immediately after every patient recruited will be evaluated with ultrasound in subcostal bicaval view
  To measure the percentage of the patients in which acoustic window is good enough to evaluate "push to bubbles" time using subcostal bicaval view.
Percentage in which "push to bubbles" time is evaluable using apical 4-chamber view | Immediately after every patient recruited will be evaluated with ultrasound in apical 4-chamber view
  To measure the percentage of the patients in which acoustic window is good enough to evaluate "push to bubbles" time using 4-chamber view.
Difference between "push to bubbles" time averages measured using the three different ultrasound views with the catheter tip in right atrium | Immediately after "push to bubbles" time will be evaluated in every patient recruited using the three different ultrasound views with the catheter tip in right atrium
  To determine if there is a significative difference between "push to bubbles" time averages measured using the three different ultrasound views: subcostal 4-chamber view, subcostal bicaval view and apical 4-chamber view with the catheter tip in right atrium
Difference between "push to bubbles" time averages measured using the three different ultrasound views with the catheter tip at the CAJ | Immediately after "push to bubbles" time will be evaluated in every patient recruited using the three different ultrasound views with the catheter tip at the CAJ
  To determine if there is a significative difference between "push to bubbles" time averages measured using the three different ultrasound views: subcostal 4-chamber view, subcostal bicaval view and apical 4-chamber view with the catheter tip at the CAJ
Difference between "push to bubbles" time averages measured using the three different ultrasound views with the catheter tip at 4 centimeters proximal to CAJ, in superior vena cava | Immediately after "push to bubbles" time will be evaluated in every patient recruited using the three different ultrasound views with the catheter tip at 4 centimeters proximal to CAJ
  To determine if there is a significative difference between "push to bubbles" time averages measured using the three different ultrasound views: subcostal 4-chamber view, subcostal bicaval view and apical 4-chamber view with the catheter tip at 4 centimeters proximal to CAJ, in superior vena cava
Difference between "push to bubbles" time averages measured using the three different ultrasound views with the catheter tip at 8 centimeters proximal to CAJ | Immediately after "push to bubbles" time will be evaluated in every patient recruited using the three different ultrasound views with the catheter tip at 8 centimeters proximal to CAJ
  To determine if there is a significative difference between "push to bubbles" time averages measured using the three different ultrasound views: subcostal 4-chamber view, subcostal bicaval view and apical 4-chamber view with the catheter tip at 8 centimeters proximal to CAJ
Evaluation of the quality of bubbles flow when the catheter tip is in the right atrium, using subcostal 4-chamber view | Immediately after Immediately after the evaluation of time for the right atrium to be completely filled by micro bubbles with the catheter tip placed in right atrium using subcostal 4-chamber view
  To evaluate the percentage in which the bubbles flow is laminar or turbulent when the catheter tip is in the right atrium, using subcostal 4-chamber view
Evaluation of the quality of bubbles flow when the catheter tip is in the right atrium, using subcostal bicaval view | Immediately after the evaluation of time for the right atrium to be completely filled by micro bubbles with the catheter tip placed in right atrium using subcostal bicaval view
  To evaluate the percentage in which the bubbles flow is laminar or turbulent when the catheter tip is in the right atrium, using subcostal bicaval view
Evaluation of the quality of bubbles flow when the catheter tip is in the right atrium, using apical 4-chamber view | Immediately after the evaluation of time for the right atrium to be completely filled by micro bubbles with the catheter tip placed in right atrium using apical 4-chamber view
  To evaluate the percentage in which the bubbles flow is laminar or turbulent when the catheter tip is in the right atrium, using apical 4-chamber view
Evaluation of the quality of bubbles flow when the catheter tip is at the CAJ using subcostal 4-chamber view | Immediately after the evaluation of time for the right atrium to be completely filled by micro bubbles with the catheter tip placed in right atrium using subcostal 4-chamber view
  To evaluate the percentage in which the bubbles flow is laminar or turbulent when the catheter tip is at the CAJ, using subcostal 4-chamber view
Evaluation of the quality of bubbles flow when the catheter tip is at the CAJ, using subcostal bicaval view | Immediately after the evaluation of time for the right atrium to be completely filled by micro bubbles with the catheter tip placed at the CAJ using subcostal bicaval view
  To evaluate the percentage in which the bubbles flow is laminar or turbulent when the catheter tip is at the CAJ, using subcostal bicaval view
Evaluation of the quality of bubbles flow when the catheter tip is at 4 centimeters proximal to CAJ, using subcostal 4-chamber view | Immediately after the evaluation of time for the right atrium to be completely filled by micro bubbles with the catheter tip placed at 4 centimeters proximal to CAJ, using subcostal 4-chamber view
  To evaluate the percentage in which the bubbles flow is laminar or turbulent when the catheter tip is at 4 centimeters proximal to CAJ, using subcostal 4-chamber view
Evaluation of the quality of bubbles flow when the catheter tip is at 4 centimeters proximal to CAJ, using subcostal bicaval view | Immediately after the evaluation of time for the right atrium to be completely filled by micro bubbles with the catheter tip placed at 4 centimeters proximal to CAJ, using subcostal bicaval view
  To evaluate the percentage in which the bubbles flow is laminar or turbulent when the catheter tip is at 4 centimeters proximal to CAJ, using subcostal bicaval view
Evaluation of the quality of bubbles flow when the catheter tip is at 4 centimeters proximal to CAJ, using subcostal apical 4-chamber view | Immediately after the evaluation of time for the right atrium to be completely filled by micro bubbles with the catheter tip placed at 4 centimeters proximal to CAJ, using subcostal apical 4-chamber view
  To evaluate the percentage in which the bubbles flow is laminar or turbulent when the catheter tip is at 4 centimeters proximal to CAJ, using subcostal apical 4-chamber view
Evaluation of the quality of bubbles flow when the catheter tip is at 8 centimeters proximal to CAJ, using subcostal 4-chamber view | Immediately after the evaluation of time for the right atrium to be completely filled by micro bubbles with the catheter tip placed at 8 centimeters proximal to CAJ, using subcostal 4-chamber view
  To evaluate the percentage in which the bubbles flow is laminar or turbulent when the catheter tip is at 8 centimeters proximal to CAJ, using subcostal 4-chamber view
Evaluation of the quality of bubbles flow when the catheter tip is at 8 centimeters proximal to CAJ, using subcostal bicaval view | Immediately after the evaluation of time for the right atrium to be completely filled by micro bubbles with the catheter tip placed at 8 centimeters proximal to CAJ, using subcostal bicaval view
  To evaluate the percentage in which the bubbles flow is laminar or turbulent when the catheter tip is at 8 centimeters proximal to CAJ, using subcostal bicaval view
Evaluation of the quality of bubbles flow when the catheter tip is at 8 centimeters proximal to CAJ, using apical 4-chamber view | Immediately after the evaluation of time for the right atrium to be completely filled by micro bubbles with the catheter tip placed at 8 centimeters proximal to CAJ, using apical 4-chamber view
  To evaluate the percentage in which the bubbles flow is laminar or turbulent when the catheter tip is at 8 centimeters proximal to CAJ, using apical 4-chamber view
Correlation between heart rate and "push to bubbles" time measured with the catheter tip placed in right atrium using subcostal 4-chamber view | Heart rate will be measured immediately before the ultrasound video recording with the catheter tip placed in right atrium using subcostal 4-chamber view
  To correlate the heart rate measured immediately before the ultrasound video recording with the catheter tip placed in right atrium using subcostal 4-chamber view
Correlation between heart rate and "push to bubbles" time measured with the catheter tip placed at CAJ using subcostal 4-chamber view | Heart rate will be measured immediately before the ultrasound video recording with the catheter tip placed at CAJ using subcostal 4-chamber view
  To correlate the heart rate measured immediately before the ultrasound video recording with the catheter tip placed at CAJ using subcostal 4-chamber view
Correlation between heart rate and "push to bubbles" time measured with the catheter tip placed at 4 centimeters proximal to CAJ, in superior vena cava, using subcostal 4-chamber view | Heart rate wil be measured immediately before the ultrasound video recording with the catheter tip placed at 4 centimeters proximal to CAJ, in superior vena cava using subcostal 4-chamber view
  To correlate the heart rate measured immediately before the ultrasound video recording with the catheter tip placed at 4 centimeters proximal to CAJ, in superior vena cava using subcostal 4-chamber view
Correlation between heart rate and "push to bubbles" time measured with the catheter tip placed at 8 centimeters proximal to CAJ, using subcostal 4-chamber view | Heart rate will be measured immediately before the ultrasound video recording with the catheter tip placed at at 8 centimeters proximal to CAJ, using subcostal 4-chamber view
  To correlate the heart rate measured immediately before the ultrasound video recording with the catheter tip placed at 8 centimeters proximal to CAJ, using subcostal 4-chamber view
Correlation between systolic arterial blood pressure and "push to bubbles" time measured with the catheter tip placed in right atrium, using subcostal 4-chamber view | Systolic arterial blood pressure will be measured immediately before the ultrasound video recording the contrast injection with the catheter tip placed in right atrium, using subcostal 4-chamber view
  To correlate the systolic arterial blood pressure measured immediately before the ultrasound video recording with the catheter tip placed in right atrium, using subcostal 4-chamber view
Correlation between systolic arterial blood pressure and "push to bubbles" time measured with the catheter tip placed at CAJ, using subcostal 4-chamber view | Systolic arterial blood arterial pressure will be measured immediately before the ultrasound video recording with the catheter tip placed at CAJ, using subcostal 4-chamber view
  To correlate the systolic arterial blood pressure measured immediately before the ultrasound video recording with the catheter tip placed at CAJ, using subcostal 4-chamber view
Correlation between systolic arterial blood pressure and "push to bubbles" time measured with the catheter tip placed at 4 centimeters proximal to CAJ, using subcostal 4-chamber view | Systolic arterial blood pressure is measured immediately before the ultrasound video recording the contrast injection with the catheter tip placed at 4 centimeters proximal to CAJ, using subcostal 4-chamber view
  To correlate the systolic arterial blood pressure recorded immediately before the ultrasound video with the catheter tip placed at 4 centimeters proximal to CAJ, using subcostal 4-chamber view
Correlation between systolic arterial blood pressure and "push to bubbles" time measured with the catheter tip placed at 8 centimeters proximal to CAJ, using subcostal 4-chamber view | Systolic arterial blood pressure is measured immediately before the ultrasound video with the catheter tip placed at 8 centimeters proximal to CAJ, using subcostal 4-chamber view
  To correlate the systolic arterial blood pressure measured immediately before the ultrasound video with the catheter tip placed at 8 centimeters proximal to CAJ, using subcostal 4-chamber view
Correlation between mean arterial blood pressure and "push to bubbles" time measured with the catheter tip placed in right atrium, using subcostal 4-chamber view | Mean arterial blood pressure is measured immediately before the ultrasound video recording with the catheter tip in right atrium, using subcostal 4-chamber view
  To correlate the mean arterial blood measured immediately before the ultrasound video recording with the catheter tip placed in right atrium, using subcostal 4-chamber view
Correlation between mean arterial blood pressure and "push to bubbles" time measured with the catheter tip placed at CAJ, using subcostal 4-chamber view | Mean arterial blood pressure is measured immediately before the ultrasound video recording with the catheter tip at CAJ, using subcostal 4-chamber view
  To correlate the mean arterial blood measured immediately before the ultrasound video recording with the catheter tip placed at CAJ, using subcostal 4-chamber view
Correlation between mean arterial blood pressure and "push to bubbles" time measured with the catheter tip placed at 4 centimeters proximal to CAJ, using subcostal 4-chamber view | Mean arterial blood pressure is measured immediately before the ultrasound video recording with the catheter tip at 4 centimeters proximal to CAJ, using subcostal 4-chamber view
  To correlate the mean arterial blood measured immediately before the ultrasound video recording with the catheter tip placed at 4 centimeters proximal to CAJ, using subcostal 4-chamber view
Correlation between mean arterial blood pressure and "push to bubbles" time measured with the catheter tip placed at 8 centimeters proximal to CAJ, using subcostal 4-chamber view | Mean arterial blood pressure is measured immediately before the ultrasound video recording with the catheter tip at 8 centimeters proximal to CAJ, using subcostal 4-chamber view
  To correlate the mean arterial blood measured immediately before the ultrasound video recording with the catheter tip placed at 8 centimeters proximal to CAJ, using subcostal 4-chamber view
Correlation between diastolic arterial blood pressure and "push to bubbles" time measured with the catheter tip placed in right atrium, using subcostal 4-chamber view | Diastolic arterial blood pressure is measured immediately before the ultrasound video recording with the catheter tip in right atrium, using subcostal 4-chamber view
  To correlate the diastolic arterial blood measured immediately before the ultrasound video recording with the catheter tip placed in right atrium using subcostal 4-chamber view
Correlation between diastolic arterial blood pressure and "push to bubbles" time measured with the catheter tip placed at CAJ, using subcostal 4-chamber view | Diastolic arterial blood pressure is measured immediately before the ultrasound video recording with the catheter tip at CAJ, using subcostal 4-chamber view
  To correlate the diastolic arterial blood measured immediately before the ultrasound video recording with the catheter tip placed at CAJ using subcostal 4-chamber view
Correlation between diastolic arterial blood pressure and "push to bubbles" time measured with the catheter tip placed at 4 centimeters proximal to CAJ, using subcostal 4-chamber view | Diastolic arterial blood pressure is measured immediately before the ultrasound video recording with the catheter tip at 4 centimeters proximal to CAJ, using subcostal 4-chamber view
  To correlate the diastolic arterial blood measured immediately before the ultrasound video recording with the catheter tip placed at 4 centimeters proximal to CAJ using subcostal 4-chamber view
Correlation between diastolic arterial blood pressure and "push to bubbles" time measured with the catheter tip placed at 8 centimeters proximal to CAJ, using subcostal 4-chamber view | Diastolic arterial blood pressure is measured immediately before the ultrasound video recording with the catheter tip at 8 centimeters proximal to CAJ, using subcostal 4-chamber view
  To correlate the diastolic arterial blood measured immediately before the ultrasound video recording with the catheter tip placed at 8 centimeters proximal to CAJ using subcostal 4-chamber view
Correlation between systolic pulmonary artery pressure and "push to bubbles" time measured with the catheter tip placed in right atrium, using subcostal 4-chamber view | Systolic pulmonary artery pressure is measured immediately before the ultrasound video recording with the catheter tip in right atrium, using subcostal 4-chamber view
  To correlate the systolic pulmonary artery pressure measured immediately before the ultrasound video recording with the catheter tip placed in right atrium, using subcostal 4-chamber view
Correlation between systolic pulmonary artery pressure and "push to bubbles" time measured with the catheter tip placed at CAJ, using subcostal 4-chamber view | Systolic pulmonary artery pressure is measured immediately before the ultrasound video recording with the catheter tip at CAJ, using subcostal 4-chamber view
  To correlate the systolic pulmonary artery pressure measured immediately before the ultrasound video recording with the catheter tip placed at CAJ, using subcostal 4-chamber view
Correlation between systolic pulmonary artery pressure and "push to bubbles" time measured with the catheter tip placed at 4 centimeters proximal to CAJ, using subcostal 4-chamber view | Systolic pulmonary artery pressure is measured immediately before the ultrasound video recording with the catheter tip at 4 centimeters proximal to CAJ, using subcostal 4-chamber view
  To correlate the systolic pulmonary artery pressure measured immediately before the ultrasound video recording with the catheter tip placed at 4 centimeters proximal to CAJ, using subcostal 4-chamber view
Correlation between systolic pulmonary artery pressure and "push to bubbles" time measured with the catheter tip placed at 8 centimeters proximal to CAJ, using subcostal 4-chamber view | Systolic pulmonary artery pressure is measured immediately before the ultrasound video recording with the catheter tip at 8 centimeters proximal to CAJ, using subcostal 4-chamber view
  To correlate the systolic pulmonary artery pressure measured immediately before the ultrasound video recording with the catheter tip placed at 8 centimeters proximal to CAJ, using subcostal 4-chamber view
Correlation between diastolic pulmonary artery pressure and "push to bubbles" time measured with the catheter tip placed in right atrium, using subcostal 4-chamber view | Diastolic pulmonary artery pressure is measured immediately before the ultrasound video recording with the catheter tip placed in right atrium, using subcostal 4-chamber view
  To correlate the diastolic pulmonary artery pressure measured immediately before the ultrasound video recording with the catheter tip placed in right atrium, using subcostal 4-chamber view
Correlation between diastolic pulmonary artery pressure and "push to bubbles" time measured with the catheter tip placed at CAJ, using subcostal 4-chamber view | Diastolic pulmonary artery pressure is measured immediately before the ultrasound video recording with the catheter tip placed at CAJ, using subcostal 4-chamber view
  To correlate the diastolic pulmonary artery pressure measured immediately before the ultrasound video recording with the catheter tip placed at CAJ, using subcostal 4-chamber view
Correlation between diastolic pulmonary artery pressure and "push to bubbles" time measured with the catheter tip placed at 4 centimeters proximal to CAJ, using subcostal 4-chamber view | Diastolic pulmonary artery pressure is measured immediately before the ultrasound video recording with the catheter tip placed at 4 centimeters proximal to CAJ, using subcostal 4-chamber view
  To correlate the diastolic pulmonary artery pressure measured immediately before the ultrasound video recording with the catheter tip placed at 4 centimeters proximal to CAJ, using subcostal 4-chamber view
Correlation between diastolic pulmonary artery pressure and "push to bubbles" time measured with the catheter tip placed at 8 centimeters proximal to CAJ, using subcostal 4-chamber view | Diastolic pulmonary artery pressure is measured immediately before the ultrasound video recording with the catheter tip placed at 8 centimeters proximal to CAJ, using subcostal 4-chamber view
  To correlate the diastolic pulmonary artery pressure measured immediately before the ultrasound video recording with the catheter tip placed at 8 centimeters proximal to CAJ, using subcostal 4-chamber view
Correlation between central venous pressure and "push to bubbles" time measured with the catheter tip placed in right atrium, using subcostal 4-chamber view | Central venous pressure is measured immediately before the ultrasound video recording with the catheter tip placed in right atrium, using subcostal 4-chamber view
  To correlate the central venous pressure measured immediately before the ultrasound video recording with the catheter placed in right atrium, using subcostal 4-chamber view
Correlation between central venous pressure and "push to bubbles" time measured with the catheter tip placed at CAJ, using subcostal 4-chamber view | Central venous pressure is measured immediately before the ultrasound video recording with the catheter tip placed at CAJ, using subcostal 4-chamber view
  To correlate the central venous pressure measured immediately before the ultrasound video recording with the catheter tip placed at CAJ, using subcostal 4-chamber view
Correlation between central venous pressure and "push to bubbles" time measured with the catheter tip placed at 4 centimeters proximal to CAJ, using subcostal 4-chamber view | Central venous pressure is measured immediately before the ultrasound video recording with the catheter tip placed at 4 centimeters proximal to CAJ, using subcostal 4-chamber view
  To correlate the central venous pressure measured immediately before the ultrasound video recording with the catheter tip placed at 4 centimeters proximal to CAJ, using subcostal 4-chamber view
Correlation between central venous pressure and "push to bubbles" time measured with the catheter tip placed at 8 centimeters proximal to CAJ, using subcostal 4-chamber view | Central venous pressure is measured immediately before the ultrasound video recording with the catheter tip placed at 8 centimeters proximal to CAJ, using subcostal 4-chamber view
  To correlate the central venous pressure measured immediately before the ultrasound video recording with the catheter tip placed at 8 centimeters proximal to CAJ, using subcostal 4-chamber view
Correlation between cardiac output and "push to bubbles" time measured with the catheter tip placed in right atrium, using subcostal 4-chamber view | Cardiac output is measured immediately before the ultrasound video recording with the catheter tip placed in right atrium, using subcostal 4-chamber view
  To correlate the cardiac output measured immediately before the ultrasound video recording with the catheter tip placed in right atrium, using subcostal 4-chamber view
Correlation between cardiac output and "push to bubbles" time measured with the catheter tip placed at CAJ, using subcostal 4-chamber view | Cardiac output is measured immediately before the ultrasound video recording with the catheter tip placed at CAJ, using subcostal 4-chamber view
  To correlate the cardiac output measured immediately before the ultrasound video recording with the catheter tip placed at CAJ, using subcostal 4-chamber view
Correlation between cardiac output and "push to bubbles" time measured with the catheter tip placed at 4 centimeters proximal to CAJ, using subcostal 4-chamber view | Cardiac output is measured immediately before the ultrasound video recording with the catheter tip placed at 4 centimeters proximal to CAJ, using subcostal 4-chamber view
  To correlate the cardiac output measured immediately before the ultrasound video recording with the catheter tip placed at 4 centimeters proximal to CAJ, using subcostal 4-chamber view
Correlation between cardiac output and "push to bubbles" time measured with the catheter tip placed at 8 centimeters proximal to CAJ, using subcostal 4-chamber view | Cardiac output is measured immediately before the ultrasound video recording with the catheter tip placed at 8 centimeters proximal to CAJ, using subcostal 4-chamber view
  To correlate the cardiac output measured immediately before the ultrasound video recording with the catheter tip placed at 8 centimeters proximal to CAJ, using subcostal 4-chamber view

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Arlotta, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Gabriella Arlotta, Roma, Italy